CLINICAL TRIAL: NCT03547505
Title: Comparison of the Incidence of Postoperative Pain After Glide Path Preparation Using Manual, Reciprocating and Continuous Rotary Instruments: A Randomized Clinical Trial
Brief Title: Incidence of Postoperative Pain After Glide Path Preparation Using Three Different Instruments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Cangül Keskin, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KAEK-357
Record Dates: First submitted 2018-05-11; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pain
Keywords: Glide path; postoperative pain; R-Pilot; ProGlider
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- R-Pilot® (Experimental): R-Pilot® was operated by an endomotor (VDW Silver, Munich, Germany) at "Reciproc All" setting.
  Interventions: Procedure: R-Pilot®
- ProGlider® (Experimental): ProGlider® was operated by an endodontic motor (X-Smart, Dentsply Sirona, Ballaigues, Switzerland) with 16:1 contra angle at the suggested settings (300 rpm on display, 5 Ncm).
  Interventions: Procedure: ProGlider®
- Manual preparation (Experimental): In the manual glide path group, glide path creation was performed with stainless steel #08, 10, 15 K-files used with "push and pull" motion. Instruments were used with a motion in which the instrument proceeds apically quarterly to the point of resistance, then is pulled out for debris removal. The procedure was repeated with each file until the working length was achieved and confirmed with an electronic apex locator (Root ZX Mini, Morita Corp., Kyoto, Japan).
  Interventions: Procedure: Manual preparation

INTERVENTIONS:
Procedure: R-Pilot® — Glide path preparation using R-Pilot® in reciprocating manner.
  Other Names: Glide path preparation; Reciprocating glide path instrument; R-Pilot, VDW, Munich, Germany
  Arms: R-Pilot®
Procedure: ProGlider® — Glide path preparation using ProGlider® in a rotating manner.
  Other Names: Rotating glide path instrument; ProGlider, Dentsply Sirona, Ballaigues, Switzerland
  Arms: ProGlider®
Procedure: Manual preparation — Glide path preparation using manual K-files numbered from 08 to 15.
  Other Names: Glide path creation with stainless steel hand files; K-files, Dentsply Sirona, Switzerland
  Arms: Manual preparation

SUMMARY:
Endodontic postoperative pain is described as a sensation of discomfort following the completion of root canal treatment and is experienced by the 25-40% of the patients regardless of pulp and periradicular diseases (1, 2). Prevalence of pain has been reported to decrease from 40% in the first 48 hours to 11% after 7 days (2). Mechanisms of endodontic postoperative pain is multifactorial and procedural processes such as glide path preparation, establishment of apical patency or root canal instrumentation technique were claimed to influence the posttreatment pain incidence (3-5).

Glide path preparation has been reported to guide the successor instruments and prevent complications of root canal preparation such as taper lock, instrument separation, transportation, and ledge formation (6-8). Several instruments and techniques have been suggested for the preparation of glide path, including hand preparation with stainless steel K-files, the combination of reciprocating handpiece and stainless steel K-files or the use of a less tapered motor-driven nickel-titanium (NiTi) rotary instrument (9-11). The use of NiTi rotary instruments has been associated with a less time-consuming and safe glide path preparation, which respects to the original canal anatomy (9, 10).

The ProGlider (Dentsply Sirona; Ballaigues, Switzerland) is a rotary glide path instrument manufactured from memory NiTi wire, which provides increased fatigue resistance, compared to the conventional NiTi glide path instruments (12). The concept of reciprocation motion was introduced with the expectation of a safer instrumentation with a single file (13). Reciprocation motion has been reported to increase the fatigue resistance of the instrument by exerting to lower stress values compared to the continuous rotation (14). The R-Pilot (VDW; Munich, Germany) instrument introduces the reciprocating motion to the glide path preparation (15). Reciprocating motion has been reported to produce greater amount of apically extruded debris, which was associated with irritation of periradicular tissues and postoperative endodontic pain, compared to continuous motion (16). However, a few clinical trials compared the reciprocation and rotation kinematics regarding their effect on postoperative pain and reported conflicting results, which could be attributed to the use of different instrumentation systems with different mechanical properties and designs (17-19). However, the effect of reciprocating motion during glide path preparation on the postoperative endodontic pain has not been investigated, yet. The purpose of the present study was to evaluate the incidence of postoperative pain after glide path preparation performed with stainless steel K-files, ProGlider or R-Pilot glide path instruments. The null hypothesis tested was that there is no difference in the incidence and severity of postoperative pain following the glide path preparation with any of the 3 instruments.

DETAILED DESCRIPTION:
For this study, ethical board approval was given by the local university clinical researches ethical committee (KAEK-357). This study included a total of 240 patients (137 women and 103 men) between the ages of 18 and 60. According to the a priori sample size calculation using G*Power software (G*Power 3.1 for Macintosh, Heinrich-Heine, Düsseldorf, Germany) and the results of a previous study (20) a minimum sample size of 66 would be required based on a type I error of 0.05 and a power of 90% to detect differences among 3 study groups at 6 measurement times. In the present study, 80 patients were assigned to each group. Maxillary and mandibular teeth of healthy patients, who were diagnosed with asymptomatic irreversible pulpitis, symptomatic irreversible pulpitis, symptomatic apical periodontitis or asymptomatic apical periodontitis, were included to the study. Patients, who were diagnosed with acute or chronic apical abscesses, showing signs of systemic infection, having allergies to local anesthetic agents, taking medication (analgesic, antibiotic or anti-inflammatory drugs) during the 7 days before the procedure, presenting with multiple teeth requiring treatment or having a progressive periodontal disease, were excluded from the study (Fig. 1). All participants were informed about the study and had signed the written informed consent prior to treatment.

Pulp vitality was tested using thermal and electric pulp tests (Parkell, NY, USA) and confirmed and recorded after access cavity preparation according to the presence of bleeding. Periapical radiographs were taken using phosphor plates and digital radiologic system (Sirona Vario DG, Bensheim, Germany) and achieved. Clinical and radiological data were recorded on each patient's sheet and analyzed by 2 blinded examiners who were experienced endodontists. In case of conflict a third opinion was taken from another endodontist. The examiners were previously calibrated by a case series evaluation and consensus between examiners was analyzed by Kappa test, until interexaminer reliability between 0.90-1.00 was expected. Baseline demographic and clinical features of each patient (pulp vitality, tooth type, presence and level of preoperative pain) were registered (Table 1).

The subjects were treated by 4 endodontists between July 2017 and April 2018. Prior to treatment the patients were instructed how to complete a visual analogue scale (VAS) to determine their pain scores. The VAS included a 10 cm straight horizontal line numbered at each centimetre from 0 to 10. Local anesthesia using 4% articaine with adrenaline 1:100.000 was performed to all patients. In case of requirement another carpule of 4% articaine was used. Following preparation of access cavity each patient was randomly assigned to 1 of the 3 experimental groups by choosing a closed envelope, which was written the group name.

In manual glide path group, glide path creation was performed with stainless steel #08, 10, 15 K-files used with "push and pull" which was described in a previous study (21). Instruments were used with a motion, which the instrument proceeds apically quarterly to the point of resistance then pulled out for debris removal. The procedure was repeated with each file until the working length (WL) was achieved and confirmed with electronic apex locator (Root ZX Mini, Morita Corp., Kyoto, Japan).

In ProGlider group, #08 stainless steel files were used to measure WL with electronic apex locator (Morita Corp., Kyoto, Japan). ProGlider instrument was operated by an endodontic motor (X-Smart, Dentsply Sirona, Ballaigues, Switzerland) with 16:1 contra angle at the suggested settings (300 rpm on display, 5 Ncm) at the measured WL.

In R-Pilot group, #08 stainless steel files were used to measure WL with electronic apex locator (Morita Corp., Kyoto, Japan). R-Pilot instrument was operated by an endomotor (VDW Silver, Munich, Germany) at "Reciproc All" setting at the measured WL.

After glide path creation, further endodontic procedures were standardized. The root canals were prepared up to X3 instrument of ProTaper Next (Dentsply Sirona) rotary instrumentation system. In case of requirement root canals were enlarged up to X4 or X5 instrument of ProTaper Next. Irrigation was performed with 5.25% NaOCl delivered with 30-G needle syringe for 10 mL for each root canal. Following preparation each root canal was flushed with 2.5 mL of 17% EDTA for 1 minute, 2.5 mL distilled water and 2.5 mL of 5.25% NaOCl, respectively as final irrigation. Root canals were dried with sterile paper points and obturated by cold lateral compaction technique using epoxy resin sealer and gutta-percha. Access cavities were restored with temporary glass ionomer filling (Riva Light Cure, Southern Dental Industries-SDI, Australia). Then the patients were discharged with VAS forms. The patients were contacted each day for 3 days for the record of their VAS score at the post operative 6th, 12th, 18th, 24th, 48th, and 72nd hours and any possible analgesic intake.

Distribution of age, gender, tooth type, presence/absence of preoperative pain and pulp vitality among the experimental groups were tested using chi-square test whereas the level of preoperative pain scores at each group was compared using one-way analysis of variance test. Kolmogorov-Smirnov test was performed to test the distribution of VAS score data and comparisons among the preparation groups regarding the severity of postoperative pain were measured by one-way analysis of variance and post-hoc Tukey tests for each measurement interval. A logistic regression analysis was performed to determine the categorical variables such as group, age (categorized according to decades), gender, tooth type (incisor, premolar, molar), presence of preoperative pain and pulp vitality that best correlated with postoperative pain incidence. All statistical analyses were performed using SPSS software (v.18.0; IBM Corp., Chicago, IL, USA) with a level of significance set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with no systemic disease or condition
* Patients having a maxillary or mandibular teeth diagnosed with one of the plural and periodontal diseases (asymptomatic irreversible pulpitis, symptomatic irreversible pulpitis, symptomatic apical periodontitis or asymptomatic apical periodontitis)

Exclusion Criteria:

* Patients, who were diagnosed with acute or chronic apical abscesses
* Patients showing signs of systemic infection
* Patients with allergies to local anesthetic agents,
* Patients who are taking medication (analgesic, antibiotic or anti-inflammatory drugs) during the 7 days before the procedure
* Patients presenting with multiple teeth requiring treatment or having a progressive periodontal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Scores using Visual Analogue Scale (VAS) | 72 hours
  VAS is a measure of pain intensity. In the present study, the VAS included a 10 cm straight horizontal line numbered at each centimetre from 0 to 10 showing two extreme symptoms of pain. "0" means no pain and "10" means the worst pain the subject has ever experienced. Each centimeter represents the pain intensity that the subject will mark orientated from 0 to 10. The intensity is increased from 0 to 10, therefore a higher score means a higher pain intensity. There are no subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No